CLINICAL TRIAL: NCT07105995
Title: Effects of Test Foods of Different Hardness and Size on Mandibular Movements and Occlusal Morphology.
Brief Title: Investigation of Test Foods With Different Hardness and Size on Lower Jaw Movements and Occlusal Morphology Which Designed With Chewing Registrations of Different Test Foods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayşenur Özcan-Sezgin, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/102 Rev1
Record Dates: First submitted 2025-07-18; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Occlusal Morphology Design With Chewing Recordings
Keywords: occlusal morphology; digital dentistry; jaw motion tracking; virtual articulator
MeSH Terms: interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Data collection (Experimental): After enrollment of each participants data collection will be started. Data collection is the only arm of the study. This study does not have any control groups of participants. There are 7 different data collection methods. Lower jaw movements and chewing cycles of each participant will be recorded with different methods and occlusal morphologies will be designed with the data collected from each method.
  After that, researchers will design occlusal morphologies with collected data and overlap the designs with participants original occlusal anatomy which obtained from intraoral scans.
  Interventions: Other: Examination and questionnaire; Other: Intraoral scanning; Other: Facebow registrations; Other: Mandibular border movement registrations; Other: Chewing registrations

INTERVENTIONS:
Other: Examination and questionnaire — Participants will be enrolled in the study and will complete the Temporomandibular Disorders/Diagnostic Criteria (TMD/DC) questionnaire. Subsequently, the investigator will conduct a clinical examination to assess each participant's eligibility based on the predefined inclusion criteria.
Other: Intraoral scanning — The investigator will perform intraoral scanning of the participants' maxillary and mandibular dentitions, as well as record the bite registration.
Other: Facebow registrations — The investigator will perform facebow registrations on the participants utilizing an optoelectronic tracking device.
Other: Mandibular border movement registrations — The investigator will perform mandibular border movement registrations utilizing an optoelectronic mandibular movement tracking device.
Other: Chewing registrations — The investigator will perform 5 chewing registrations with different test foods utilizing an optoelectronic mandibular movement tracking device.

SUMMARY:
One of the most important goals of prosthetic treatment is to make the occlusal morphology suitable for the patient's original anatomy. Mechanical articulators are metal devices that mimic the temporomandibular joint and lower jaw movements, and attempts have been made to make them patient-specific over the years. For this purpose, semi-adjustable articulators were first developed. Later, fully adjustable articulators were introduced to the market. Although these devices have the closest imitation mechanism to the patient's original anatomy, they have various limitations. Adjusting mechanical articulators and recording lower jaw movements have been researched in dentistry clinics and dentistry literature for many years. Due to the limitations of articulators, digital recordings of lower jaw movements have been started since 1989. Later, in 2002, the process of adjusting virtual articulators in a computer environment according to the digital recording data of the mandibular movements was started. In this way, the limitations of mechanical articulators such as metal deformation, difficulties experienced during recording, distortion of plaster and recording material, insufficient stability, adaptation problems of base plates, logistic problems between the laboratory and the physician, and inability to store data have been largely eliminated. In addition, mechanical articulators still cannot fully mimic the anatomy of the temporomandibular joint and related muscles. Digital recording of mandibular movements and transferring them to a virtual environment were first tried with electronic methods, and these systems were developed and ultrasonic and optoelectronic methods were used. Today, tooth movement records can be obtained with 3D video motion analysis methods. By superimposing these data with the data of digital models of the jaws, a mandibular movement recording method has been developed that can now produce restorations without the need for virtual or mechanical articulators. All these developments arise from the desire to record more appropriate and adaptable mandibular movement patterns, overcoming the difficulties in imitating complex patterns of mandibular movements that vary from the size, initial height and consistency of the food to the patient's mental state during the mandibular chewing movement. Thus, we will be able to obtain the most appropriate occlusal morphology for the patient to chew at maximum performance in the prosthetic or restorative procedures we will perform. With the developing technology, mandibular movement recordings can be recorded not only in the border movements as in the past, but also during chewing. In the literature, the majority of studies conducted by having the patient chew a test food are studies measuring the activity of the masticatory muscles, the distance between the incisors, the lateral movement distance or the magnitude of the chewing stroke.

For this reason, in this study, mandibular movements will be recorded with optical motion tracking systems and 4-unit fixed partial dentures(FPDs) for teeth 4.4 - 4.7 will be designed according the recordings.

The study will include individuals who are in the molar class 1 of the Angle classification, who have no temporomandibular joint and masticatory muscle disorders, who have no missing or extra teeth, who have no fillings or crowns on teeth numbered 4.4-4.7, who have not undergone orthodontics, and who are not allergic to the test foods. The subjects will sign a consent form. After the subjects are examined, lower and upper jaw scans and bite scans will be recorded. In the 2nd session, facebow records, border movements and chewing records with 5 different test foods will be recorded from the subjects with an optical lower jaw movement tracker(Zebris JMA Optic). These test foods were selected according to the literature and are cheese, raw carrots, boiled carrots, crispy bread and pre-polymerized silicone impression material. After recordings, fixed partial dentures will be designed via virtual articulator, border movement recordings and for 5 different foods in digital design program. 7 different FDPs designs for each subject will be overlapped with the subject's original anatomy in the Geomagic program.

DETAILED DESCRIPTION:
A fundamental objective in prosthodontic rehabilitation is the accurate replication of the patient's native occlusal architecture. Since the early 20th century, dentistry has endeavored to simulate the functional dynamics of the temporomandibular joint (TMJ) and mandibular motion through the use of mechanical articulators-metallic devices engineered to replicate mandibular kinematics. Over time, these articulators have evolved from basic models to more sophisticated, patient-specific systems. Initially, semi-adjustable articulators emerged, followed by the development of fully adjustable variants intended to more closely approximate individual anatomical parameters. Despite their improved accuracy, these devices are not without limitations.

While fully adjustable articulators represent the most anatomically faithful mechanical approximation of mandibular function, they remain inherently limited in precision and adaptability. The calibration of these devices and the accurate documentation of mandibular movements have been subjects of long-standing investigation within both clinical and academic domains of dentistry. In response to the intrinsic shortcomings of mechanical systems-such as susceptibility to material deformation and challenges in capturing dynamic motion-digital motion capture technologies began to emerge in 1989. This transition marked a significant shift toward enhancing the fidelity of mandibular movement analysis.

By 2002, advancements in digital dentistry enabled the integration of virtual articulators within computer-aided design environments, utilizing digitally captured mandibular movement data. This innovation substantially addressed the limitations associated with traditional mechanical articulators, including structural deformation, inaccuracies during physical registration, degradation of plaster or recording media, and logistical inefficiencies in transferring physical components between clinical and laboratory settings. Furthermore, digital systems introduced the critical advantage of data preservation and reproducibility-parameters difficult to achieve with analog models.

Despite ongoing enhancements, mechanical articulators remain incapable of fully replicating the complex anatomical and neuromuscular intricacies of the temporomandibular joint and its associated musculature. Initial efforts to digitally capture mandibular motion involved rudimentary electronic methodologies, which were subsequently refined through the application of ultrasonic and optoelectronic tracking technologies. These innovations significantly improved the spatial resolution and reliability of movement data, enabling more sophisticated integration with virtual modeling systems.

Contemporary techniques now permit the acquisition of mandibular motion data through three-dimensional video-based motion capture systems. When these dynamic recordings are overlaid onto digitized jaw models, a new paradigm in prosthetic design is achieved-allowing for the fabrication of dental restorations without reliance on either virtual or physical articulators. This method not only enhances anatomical precision but also minimizes procedural constraints associated with traditional systems.

These advancements stem from an ongoing pursuit to capture mandibular movements with greater anatomical accuracy and functional adaptability. The inherent complexity of mandibular kinematics-modulated by factors such as food size, texture, and initial occlusal positioning, as well as psychosocial influences during mastication-has historically challenged the capacity of both clinicians and devices to simulate real-world chewing behavior. Digital methodologies offer a more nuanced and individualized representation of these dynamic patterns.

As a result, clinicians are increasingly capable of designing restorations that optimize occlusal morphology, thereby supporting maximal masticatory efficiency in prosthetic and restorative procedures. Technological advancements have expanded the scope of mandibular motion analysis beyond conventional border movements to include real-time recordings captured during functional activities such as chewing. This progression offers a more accurate representation of intraoral dynamics under natural physiological conditions.

The existing body of literature predominantly focuses on the evaluation of masticatory parameters during test food consumption, including electromyographic activity of masticatory muscles, incisal separation distances, lateral excursion amplitudes, and the overall range of chewing cycles. These studies have collectively established that mastication is highly sensitive to the physical properties of food, particularly in relation to its texture, hardness, and size.

It has been well-documented that the nature of food significantly influences mandibular kinematics, with textural variations playing a pivotal role in altering chewing patterns. Numerous studies have investigated how differences in food hardness and dimensional properties affect masticatory behavior, shedding light on the adaptive responses of the jaw during functional loading.

Findings from research examining the influence of food size on mandibular motion generally indicate a positive correlation between food volume and chewing cycle duration. As food size increases, both the intensity of masticatory muscle activation and the amplitude and velocity of mandibular movement tend to rise correspondingly-suggesting a coordinated neuromuscular adaptation to mechanical demands.

With respect to food hardness, there is broad agreement that greater hardness elicits elevated masticatory muscle activity. However, the impact of hardness on other kinematic parameters-such as cycle duration, movement amplitude, and speed-remains inconclusive, reflecting interindividual variability and methodological differences across studies.

Furthermore, the current literature lacks clinical investigations directly comparing the occlusal morphology of prosthetic restorations derived from dynamic chewing records with those fabricated through conventional mechanical or virtual articulator-based methods, including those relying solely on border movement data. This absence underscores a significant knowledge gap regarding the potential functional advantages of mastication-based modeling over traditional techniques.

To address this deficiency, the present study will utilize optoelectronic motion capture systems to record mandibular movements within the Department of Prosthodontics. The study is grounded in the following hypotheses:

Null Hypothesis (H₀):

Variations in the hardness and consistency of test foods do not induce statistically significant angular deviations in mandibular movement patterns.

Alternative Hypotheses:

H₁: Prosthetic restorations designed using functional chewing records do not exhibit differences in occlusal morphology compared to those created via conventional or virtual articulators.

H₂: Patient-specific anatomical parameters-such as condylar path inclination and the Bennett angle-remain consistent across chewing recordings conducted with various test foods.

A statistical power analysis was conducted using G*Power version 3.1.9.7 (Franz Faul, Universität Kiel, Germany), referencing the methodological parameters established in Muric's 2018 study titled "Comparing the Precision of Reproducibility of Computer-Aided Occlusal Design to Conventional Methods." An effect size of 0.25 was applied, with a Type I error rate (α) of 0.20 and a statistical power (1-β) of 80%, resulting in a calculated minimum sample size of 20 participants. To ensure sufficient representation and allow for potential attrition, the final sample size was determined to be 24 individuals. Group comparisons will be analyzed using the Kruskal-Wallis test, while the Mann-Whitney U test will be applied for post hoc pairwise comparisons.

Participants will be recruited from among volunteer students enrolled at the Faculty of Dentistry, Istanbul University. Eligible subjects who meet the inclusion criteria will be identified and registered through the Prosthodontics Clinic. Appointment scheduling will be coordinated jointly with each participant, and subsequent communication will be maintained via telephone. Given the requirement for multiple sessions per participant, ease of accessibility is a key consideration in subject selection.

Since the experimental protocol necessitates the accurate performance of mandibular movements-including laterotrusion, retrusion, and protrusion-participants familiar with these movements are preferred. Accordingly, dental students from Istanbul University, who are both knowledgeable in these functional motions and readily accessible for repeated sessions, have been selected as the study population.

To minimize confounding variables arising from individual anatomical or functional variability, only systemically and dentally healthy individuals will be included. The inclusion criteria are as follows: absence of temporomandibular joint (TMJ) disorders or masticatory muscle dysfunction; no history of orthodontic treatment; intact permanent dentition with Angle Class I molar occlusion (excluding third molars); absence of dental implants, supernumerary teeth, or extensive prosthetic restorations; and no reported orofacial pain or muscle sensitivity. Additionally, participants must not exhibit any allergies or sensitivities to the test foods, and individuals unfamiliar with the selected food items will be excluded to avoid variability due to novelty effects.

The precise execution of mandibular movements during data acquisition is essential, as these recordings directly influence the accuracy and validity of experimental outcomes. In alignment with precedent set by similar research, dental students are often selected as participants due to their familiarity with standard mandibular movement patterns and their ability to follow clinical instructions with consistency. Moreover, their typical age range (18-25 years) aligns well with the study's inclusion criteria, which specify the presence of fully erupted dentition, Angle Class I occlusion, absence of extensive restorations, and no prior prosthetic or orthodontic intervention.

Each participant was assigned a unique identification number ranging from 1 to 24, which was used consistently throughout the study for confidentiality and data tracking purposes. Prior to participation, all subjects were thoroughly informed about the study's objectives, procedures, and potential risks. Informed consent was obtained in writing, confirming their voluntary agreement to participate. Clinical examination of all subjects included the administration of the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) developed by Schiffman et al., to ensure the absence of TMJ-related pathology.

Initially, digital impressions of each participant's maxillary and mandibular arches, along with occlusal bite registrations, will be obtained using the Alliedstar intraoral scanner. The acquired datasets will be exported in Standard Tessellation Language (STL) format, enabling the creation of precise digital models for subsequent analysis and design procedures.

Subsequently, mandibular border movements will be documented using the JMA Optic optoelectronic motion capture system (Zebris GmbH, Isny, Germany). The apparatus comprises a head-mounted sensor array and a bite fork affixed to the vestibular surfaces of the mandibular teeth using autopolymerizing acrylic resin (Temdent Temporary Crown and Bridge Acrylic, Schütz Dental GmbH, Rosbach, Germany). This fixation ensures stable signal transmission without impeding mandibular closure. The bite fork is adjusted for proper leveling and retention before being secured in place.

Following acquisition of the facebow registration, the "Border Movement" module within the WinJaw 10.06 software (Zebris GmbH, Isny, Germany) will be activated on a Windows-based workstation. Subject-specific information will be entered into the system, after which the recording of mandibular border movements will commence. Participants will be instructed to perform three repetitions of each predefined mandibular movement-protrusion, retrusion, right laterotrusion, and left laterotrusion-in accordance with the manufacturer's guidelines.

Upon completion of the border movement recordings, participants will be asked to sequentially masticate five standardized test foods exhibiting varying levels of hardness and consistency. Each chewing session will be recorded using the same JMA Optic device under the "Chewing" module of the WinJaw software. These recordings will capture functional mandibular kinematics during real-time mastication for each food item, facilitating a direct comparison of motion dynamics across different material properties.

The test foods selected for this study encompass a spectrum of textural and hardness profiles:

1. Soft cheese (Sütaş Dairy Products, Istanbul, Turkey), similar texture to Gouda;
2. Raw carrots (hard texture);
3. Boiled carrots (20 minutes of boiling in boiling water, moderately soft);
4. Crispy bread (UNO Kruton, Istanbul, Turkey);
5. Pre-polymerized silicone impression material, used as a substitute for peanuts due to allergy concerns, as approved by the ethics committee. (extremely hard texture, pre-polymerized according to manufacturer's manual)

Each sample will be standardized to dimensions of 10 mm × 10 mm × 10 mm to ensure uniformity in mastication parameters.

Preparation and portioning of all test foods will be conducted under controlled conditions in the Department of Prosthodontics' designated laboratory kitchen. To maintain consistency, stainless steel molds in the form of rectangular prisms (10 × 10 × 10 mm) will be fabricated and used to shape each food sample to identical size specifications. This standardization is critical to eliminating volumetric variability during mastication analysis.

For the chewing motion analysis, the JMA Optic system will be configured via the "Chewing" module in the WinJaw software. As with prior recordings, the sensor fork will be secured to the vestibular surfaces of the mandibular dentition using acrylic resin. Participants will be instructed to chew each food sample for a standardized duration of 20 seconds. The kinematic data from each session will be recorded independently, thereby generating five distinct datasets-corresponding to the five different test foods-that will form Groups 3 through 7 in the final analysis.

Upon completion of all motion and chewing recordings, the digital maxillary and mandibular models of each participant will be imported into the Exocad 3.1 Plovdiv software suite (Exocad GmbH, Darmstadt, Germany). Utilizing the "Wax-up" module, the occlusal and incisal surfaces of the mandibular dentition will be uniformly reduced by approximately 2 millimeters to simulate tooth preparation and establish a baseline for prosthetic occlusal morphology design. This digital modification facilitates the subsequent restorative modeling phase.

Subsequent to model preparation, study cohorts will be established based on the type of mandibular movement data integrated into the design process:

Group 1: Digital models coupled with closure registration data will be mounted on a semi-adjustable virtual articulator (Artex CR, Aman Girrbach, Koblach, Austria) within the design software. Prosthetic restorations will be fabricated using this conventional virtual articulation method.

Group 2: The digital jaw models will be incorporated alongside the optoelectronically recorded border movement trajectories. This dataset will guide the design of prosthetic restorations that account for patient-specific mandibular border kinematics.

Groups 3 to 7: The digital models will be integrated with chewing movement datasets obtained from the five distinct test foods independently. Each chewing dataset will be employed to inform the occlusal morphology design, resulting in five separate restoration designs reflecting functional adaptations to varied masticatory conditions.

The finalized prosthetic occlusal designs will be exported to Geomagic Control X software (3D Systems, Rock Hill, SC, USA) for comprehensive three-dimensional superimposition analysis. This process will quantify linear and angular deviations among the various restoration groups as well as discrepancies relative to the baseline intraoral scans. The software will facilitate precise measurement of spatial differences to assess the fidelity and variability induced by differing mandibular motion inputs.

Furthermore, patient-specific anatomical parameters-such as condylar path inclinations during protrusive movement and Bennett angle metrics-extracted from device-generated reports will be systematically compared across chewing and border movement datasets to evaluate consistency and accuracy.

All statistical analyses will be performed utilizing SPSS version 28.1 (IBM Corp., Armonk, NY, USA). Prior to inferential testing, data distributions will be examined for normality employing the Kolmogorov-Smirnov test. Continuous variables will be summarized as means with standard deviations, whereas categorical variables will be presented as frequencies and percentages.

To assess the agreement between measurement methods, the mean measurement errors for each reference distance will be computed. These will subsequently be evaluated using Bland-Altman plots, appropriate for multiple observations per subject, to visualize and quantify bias and limits of agreement.

For parametric data conforming to normal distribution, group comparisons involving more than two cohorts will be conducted via one-way Analysis of Variance (ANOVA), followed by Tukey's Honestly Significant Difference (HSD) post hoc tests for pairwise group analyses.

Conversely, non-parametric data failing to meet normality assumptions will be compared using the Kruskal-Wallis test for multi-group comparisons. Where significant differences arise, Mann-Whitney U tests will be employed for post hoc pairwise evaluations. To account for multiple testing and control type I error rates, Bonferroni correction will be applied to all post hoc analyses.

A significance threshold will be set at p < 0.05 for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* having Angle molar class 1 occlusion
* over 18 years old
* not undergone any orthodontic treatment
* not having any temporomandibular or masticatory disorders
* not having any pain or sensitivity on temporomandibular joint, masticatory muscle
* not having missing teeth or implant-supported restorations
* not having fillings or crowns on teeth 4.4 - 4.7
* not having supernumerary teeth
* not allergic to test foods
* volunteering to participate
* being a student at Istanbul University Faculty of Dentistry

Exclusion Criteria:

* not having Angle molar class 1 occlusion
* under 18 years old
* undergone any orthodontic treatment
* having any temporomandibular or masticatory disorders
* having any pain or sensitivity on temporomandibular joint, masticatory muscle
* having missing teeth or implant-supported restorations
* having fillings or crowns on teeth 4.4 - 4.7
* having supernumerary teeth
* allergic to test foods
* not volunteering to participate
* not being a student at Istanbul University Faculty of Dentistry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Linear deviation of reference points on occlusal morphology | From enrollment to data collection at 12 weeks. Occlusal morphology designs will be held on design program after data collection. Participiants do not take place at this phase of the study.
  Following the superimposition of the designed occlusal morphologies onto the participants' original occlusal anatomy, thirteen reference points will be assessed for linear deviations measured in micrometers.
Angular deviation of reference points on designed occlusal morphology | From enrollment to data collection at 12 weeks. Occlusal morphology designs will be held on design program after data collection. Participiants do not take place at this phase of the study.
  Following the superimposition of the designed occlusal morphologies onto the participants' original occlusal anatomy, thirteen reference points will be assessed for angular deviations measured in micrometers."

SECONDARY OUTCOMES:
Chewing cycles amplitude | From enrollment to data collection at 12 weeks. After data collection participants do not take place on designing and analyzing phases.
  The optical jaw tracking device will record the chewing cycles of each participant. Upon completion of data acquisition, individual chewing cycles associated with each test food will be analyzed. Variations in cycle amplitude will be assessed in relation to the differing hardness and texture of the test foods. All measurements will be expressed in millimeters.
Chewing cycles width | From enrollment to data collection at 12 weeks. Occlusal morphology designs will be held on design program after data collection. Participiants do not take place at this phase of the study.
  The optical jaw tracking device will record the chewing cycles of each participant. Upon completion of data acquisition, individual chewing cycles associated with each test food will be analyzed. Variations in cycle width will be assessed in relation to the differing hardness and texture of the test foods. All measurements will be expressed in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Tonguç Sülün, PhD, Study Chair — Istanbul University
Locations (1):
- Istanbul University Department of Prosthodontics, Istanbul, Süleymaniye Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koch GK, Gallucci GO, Lee SJ. Accuracy in the digital workflow: From data acquisition to the digitally milled cast. J Prosthet Dent. 2016 Jun;115(6):749-54. doi: 10.1016/j.prosdent.2015.12.004. Epub 2016 Jan 21. PMID 26803173
- [Background] Kiseri B, Dayan SC, Yildiz M, Sulun T. The correlation between direction and amount of retrusive movement and condyle position and joint space. Cranio. 2018 Jul;36(4):250-256. doi: 10.1080/08869634.2017.1333219. Epub 2017 Jun 3. PMID 28578614
- [Background] Kohyama K, Sasaki T, Hayakawa F. Characterization of food physical properties by the mastication parameters measured by electromyography of the jaw-closing muscles and mandibular kinematics in young adults. Biosci Biotechnol Biochem. 2008 Jul;72(7):1690-5. doi: 10.1271/bbb.70769. Epub 2008 Jul 7. PMID 18603809
- [Background] Kohyama K, Mioche L, Bourdiol P. Influence of age and dental status on chewing behaviour studied by EMG recordings during consumption of various food samples. Gerodontology. 2003 Jul;20(1):15-23. doi: 10.1111/j.1741-2358.2003.00015.x. PMID 12926747
- [Background] Strozyk P, Balchanowski J. Application of numerical simulation studies to determine dynamic loads acting on the human masticatory system during unilateral chewing of selected foods. Front Bioeng Biotechnol. 2023 May 11;11:993274. doi: 10.3389/fbioe.2023.993274. eCollection 2023. PMID 37251568
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Bhatka R, Throckmorton GS, Wintergerst AM, Hutchins B, Buschang PH. Bolus size and unilateral chewing cycle kinematics. Arch Oral Biol. 2004 Jul;49(7):559-66. doi: 10.1016/j.archoralbio.2004.01.014. PMID 15126137
- [Background] Peyron MA, Lassauzay C, Woda A. Effects of increased hardness on jaw movement and muscle activity during chewing of visco-elastic model foods. Exp Brain Res. 2002 Jan;142(1):41-51. doi: 10.1007/s00221-001-0916-5. Epub 2001 Nov 9. PMID 11797083
- [Background] Cheong CW, Radomski K, Otten J, Lee SJ. A clinical comparative analysis using an optical tracking device versus conventional tracking device in the production of occlusal appliances. J Prosthodont. 2025 Apr;34(4):350-356. doi: 10.1111/jopr.13989. Epub 2024 Dec 4. PMID 39632348
- [Background] Nigam AA, Lee JD, Lee SJ. A clinical comparison of sagittal condylar inclination and Bennett angle derived from a conventional electronic tracking device and an optical jaw tracking device. J Prosthet Dent. 2025 Aug;134(2):393-398. doi: 10.1016/j.prosdent.2023.10.034. Epub 2023 Nov 28. PMID 38030543
- [Background] Muric A, Gokcen Rohlig B, Ongul D, Evlioglu G. Comparing the precision of reproducibility of computer-aided occlusal design to conventional methods. J Prosthodont Res. 2019 Jan;63(1):110-114. doi: 10.1016/j.jpor.2018.10.002. Epub 2018 Nov 13. PMID 30446412
- [Background] Lepidi L, Galli M, Mastrangelo F, Venezia P, Joda T, Wang HL, Li J. Virtual Articulators and Virtual Mounting Procedures: Where Do We Stand? J Prosthodont. 2021 Jan;30(1):24-35. doi: 10.1111/jopr.13240. Epub 2020 Sep 2. PMID 32827222
- [Background] Anderson K, Throckmorton GS, Buschang PH, Hayasaki H. The effects of bolus hardness on masticatory kinematics. J Oral Rehabil. 2002 Jul;29(7):689-96. doi: 10.1046/j.1365-2842.2002.00862.x. PMID 12153460
- [Background] Shiga H, Stohler CS, Kobayashi Y. The effect of bolus size on the chewing cycle in humans. Odontology. 2001 Nov;89(1):49-53. doi: 10.1007/s10266-001-8185-0. PMID 14530922
- [Background] Miyawaki S, Ohkochi N, Kawakami T, Sugimura M. Effect of food size on the movement of the mandibular first molars and condyles during deliberate unilateral mastication in humans. J Dent Res. 2000 Jul;79(7):1525-31. doi: 10.1177/00220345000790071601. PMID 11005739